CLINICAL TRIAL: NCT01104415
Title: A Phase 2, Open-Label, Multi-Center, Serial Ascending-Dose, Dose-Finding Study to Evaluate the Safety and Tolerability of LX1606 in Subjects With Symptomatic Carcinoid Syndrome
Brief Title: Study of Telotristat Etiprate (LX1606) in Participants With Symptomatic Carcinoid Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-203-CS; LX1606.203, LX1032 (Other: Lexicon Pharmaceuticals, Inc.); 2009-016973-13 (EudraCT Number)
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome | interventions — telotristat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telotristat etiprate - Core Phase (Experimental): Following a 2-week Run-In Period, participants received telotristat etiprate capsules at a starting dose of 150 mg, orally three times daily (TID) for 14 days in the Core Phase. Dose escalations (250 mg, 350 mg, 500 mg) occurred serially every 14 days, up to a maximum dosage of telotristat etiprate 500 mg TID, as guided by specific clinical criteria for dose escalation. Upon completion of 12 weeks of treatment, participants were eligible to receive telotristat etiprate in the optional Open-label Extension Period.
  Interventions: Drug: Telotristat etiprate
- Telotristat etiprate - Extension Period (Experimental): Participants received telotristat etiprate at their highest tolerated dose (250 mg or 500 mg), orally, TID for 124 weeks in the Open-label Extension Period. If neither dose was tolerated participants were discontinued from the study and completed the 2-week Follow-up Visit.
  Interventions: Drug: Telotristat etiprate

INTERVENTIONS:
Drug: Telotristat etiprate — Telotristat etiprate capsules orally three times daily.
  Other Names: LX1606 Hippurate

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of orally administered telotristat etiprate (LX1606) in participants with symptomatic carcinoid syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 18 and older
* Biopsy-proven metastatic carcinoid tumor of the gastrointestinal (GI) tract with disease extent confirmed by computed tomography (CT), magnetic resonance imaging (MRI), or radionuclide imaging
* Symptomatic carcinoid syndrome (≥4 bowel movements per day)
* Ability to provide written informed consent

Exclusion Criteria:

* ≥ 12 high-volume, watery bowel movements per day
* Sponsor-unacceptable clinical laboratory values for hematology and liver function tests at screening
* Karnofsky status ≤70% - unable to care for self
* Surgery within 60 days prior to screening
* A history of short bowel syndrome
* Life expectancy < 12 months
* History of substance or alcohol abuse within 2 years prior to screening
* Administration of any investigational drug within 30 days of screening or any therapeutic protein or antibody within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2014-02-12 (Actual); Study Completion 2014-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo LaPuerta, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (10):
- Germany (6):
  - Lexicon Investigational Site, Bad Berka
  - Lexicon Investigational Site, Berlin
  - Lexicon Investigational Site, Halle
  - Lexicon Investigational Site, Lübeck
  - Lexicon Investigational Site, Marburg
  - Lexicon Investigational Site, Munich
- United Kingdom (4):
  - Lexicon Investigational Site, Basingstoke
  - Lexicon Investigational Site, Cambridge
  - Lexicon Investigational Site, London
  - Lexicon Investigational Site, Manchester

REFERENCES:
- [Derived] Pavel M, Horsch D, Caplin M, Ramage J, Seufferlein T, Valle J, Banks P, Lapuerta P, Sands A, Zambrowicz B, Fleming D, Wiedenmann B. Telotristat etiprate for carcinoid syndrome: a single-arm, multicenter trial. J Clin Endocrinol Metab. 2015 Apr;100(4):1511-9. doi: 10.1210/jc.2014-2247. Epub 2015 Jan 30. PMID 25636046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 participants were enrolled in the Core Phase (8-week Dose-escalation Period and the 4-week Stable-dose Period) from 11 sites in the United Kingdom and Germany, and 11 participants entered the Open-label Extension Period.
Groups:
- Telotristat Etiprate- Core Phase: Following a 2-week Run-In Period, participants received telotristat etiprate capsules at a starting dose of 150 mg, orally three times daily (TID) for 14 days in the Core Phase. Dose escalations (250 mg, 350 mg, 500 mg) occurred serially every 14 days, up to a maximum dosage of telotristat etiprate 500 mg TID, as guided by specific clinical criteria for dose escalation. Upon completion of 12 weeks of treatment, participants were eligible to receive telotristat etiprate in the optional Open-label Extension Period.
- Telotristat Etiprate -Extension Period: Participants received telotristat etiprate at their highest tolerated dose (250 mg or 500 mg), orally, TID for 124 weeks in the Open-label Extension Period. If neither dose was tolerated participants were discontinued from the study and completed the 2-week Follow-up Visit.
Period: Core Phase
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate -Extension Period
Started | 15 | 0
Completed | 14 | 0
Not Completed | 1 | 0
Not completed — Consent withdrawn by subjects | 1 | 0
Period: Extension Period
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate -Extension Period
Started | 0 | 11 (Out of 14 participants who completed Core Phase, 3 were not eligible to enter the Extension Period.)
Completed | 0 | 0
Not Completed | 0 | 11
Not completed — Progressive disease | 0 | 4
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Transition to Study LX1606.302 | 0 | 4
Not completed — Heart surgery/feeling miserable | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all the enrolled participants who received at least 1 dose of study drug.
Arm/Group | Telotristat Etiprate- Core Phase
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6
  Germany | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment Emergent Adverse Events (TEAEs) and Drug-Related TEAEs in the Core Phase
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. Treatment-emergent AEs were defined as any AEs reported after the first dose of treatment on Day 1.
Time Frame: Baseline up to Week 12 in the Core Phase
Population: The safety set (SS) included all the enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Telotristat Etiprate- Core Phase
Number analyzed (Participants) | 15
Participants
  Any TEAE | 15
  Drug-Related TEAE | 5

2. Primary Outcome: Number of Participants With Any Treatment Emergent Adverse Events (TEAEs) and Drug-Related TEAEs in the Extension Period
Description: as for outcome 1
Time Frame: Up to 124 Weeks in the Extension Period
Population: SS included all enrolled participants who had received at least 1 dose of study drug in the 124-week Extension Period.
Measure: Count of Participants; unit: Participants
Groups:
- Telotristat Etiprate- Extension Period: Participants received telotristat etiprate at their highest tolerated dose (250 mg or 500 mg), orally, TID for 124 weeks in the Open-label Extension Period. If neither dose was tolerated participants were discontinued from the study and completed the 2-week Follow-up Visit.
Arm/Group | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 11
Participants
  Any TEAE | 11
  Drug-Related TEAE | 4

3. Secondary Outcome: Change From Baseline in Number of Bowel Movements (BMs)
Description: Participants recorded the number of bowel movements in a daily diary. The change from baseline value was calculated as the difference between mean numbers of BMs of the post-baseline interval (Weeks 9 to 12) and baseline. A negative change from baseline indicates improvement. Baseline for the Extension Period was defined as non-missing assessment in Run-in period prior to the first dose of study drug.
Time Frame: Core Phase: Baseline to Weeks 9-12; Extension Period: Baseline to Week 24
Population: Efficacy full analysis set (EFAS) in Core Phase included all participants with at least 1 post-Baseline efficacy assessment and full analysis set (FAS) in Extension Period(EP) included all participants in SS with at least 1 post-Baseline efficacy assessment in 124-week EP. Number analyzed is the participants with evaluable data at given time point.
Measure: Mean (Standard Deviation); unit: number of bowel movements/day
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 14 | 8
number of bowel movements/day | -2.60 (1.381) | -2.85 (1.64)

4. Secondary Outcome: Change From Baseline in Stool Form/Consistency
Description: Participants assessed stool form/consistency in a daily diary using a 6-point scale (0-none, 1-hard, 2-firm, 3-soft, 4-loose, 5-watery). The change from the baseline value was calculated as the difference between a mean score of the post-baseline interval (Weeks 9 to 12) and baseline. 0 indicates the best score and 5 indicates the worst score. A negative change from baseline indicates improvement. Baseline for the Extension Period was defined as non-missing assessment in Run-in period prior to the first dose of study drug.
Time Frame: Core Phase: Baseline to Weeks 9-12; Extension Period: Baseline to Week 24
Population: EFAS in the Core Phase included all participants who had at least 1 post-Baseline efficacy assessment and FAS in the Extension period included all participants in the safety set who had at least 1 post-Baseline efficacy assessment in 124-week Extension Period. Number analyzed is the number of participants with evaluable data at given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 14 | 8
score on a scale | -0.79 (0.707) | -1.31 (0.666)

5. Secondary Outcome: Change From Baseline in Percentage of Days With Sensation of Urgency to Defecate
Description: Participants assessed the urgency to defecate using a daily diary response to the following question, "Have you felt or experienced a sense of urgency to pass stool today?". The change from the baseline value was calculated as the difference between the mean score (percentage of days) of the post-baseline interval (Weeks 9 to 12) and baseline. Baseline for the Extension Period was defined as non-missing assessment in Run-in period prior to the first dose of study drug.
Time Frame: Core Phase: Baseline to Weeks 9-12; Extension Period: Baseline to Week 24
Population: EFAS in Core Phase included all participants who had at least 1 post-Baseline efficacy assessment and FAS in Extension Period included all participants in the safety set who had at least 1 post-Baseline efficacy assessment in the 124-week Extension Period. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 14 | 8
percentage of days | -11.32 (36.660) | -22.79 (49.546)

6. Secondary Outcome: Change From Baseline in Sensation/Severity of Nausea Using 100 mm Visual Analog Scale (VAS)
Description: Sensation/severity of nausea was measured using a 100 mm VAS. Participants rated their perception of the sensation/severity of nausea experienced by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No vomiting and 100 = vomiting. The change from the baseline value was calculated as the difference between the mean score of the post-baseline interval (Weeks 9 to 12) and baseline. 0 indicates the best score, 100 indicates the worst score. Baseline for the Extension Period was defined as non-missing assessment in Run-in period prior to the first dose of study drug.
Time Frame: Core Phase: Baseline to Weeks 9-12; Extension Period: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 13 | 7
score on a scale | -2.43 (5.208) | -5.71 (8.797)

7. Secondary Outcome: Number of Participants With an Improvement in Global Assessment of Symptoms Associated With Carcinoid Syndrome
Description: Participants assessed their symptoms using a weekly subjective response to the following question, "In the past 7 days, have you had adequate relief of your carcinoid syndrome bowel complaints such as diarrhea, urgent need to have a bowel movement, abdominal pain, or discomfort?". The values for improvement in global assessment of symptoms associated with carcinoid syndrome in the Core Phase were averaged from Weeks 9 to 12.
Time Frame: Core Phase: Weeks 9-12; Extension Period: Week 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 13 | 7
Participants | 10 | 4

8. Secondary Outcome: Change From Baseline in Daily Severity of Abdominal Pain or Discomfort Using 100 mm Visual Analog Scale (VAS)
Description: The severity of abdominal pain was measured using a 100 mm VAS. Participants rated their perception of the sensation/severity of abdominal pain or experienced by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No vomiting and 100 = vomiting. The change from the baseline value was calculated as the difference between the mean score of the post-baseline interval (Weeks 9 to 12) and baseline. 0 indicate the best score, 100 indicates the worst score. Baseline for the Extension Period was defined as non-missing assessment in Run-in period prior to the first dose of study drug.
Time Frame: Core Phase: Baseline to Weeks 9-12; Extension Period: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 14 | 7
score on a scale | -8.66 (18.724) | -24.11 (19.643)

9. Secondary Outcome: Change From Baseline in Daily Number of Cutaneous Flushing Episodes
Description: Participants recorded the number of daily cutaneous flushing episodes experienced in the daily diary. The change from baseline value was calculated as the difference between the mean numbers of cutaneous flushing episodes of the post-baseline interval (Weeks 9 to 12) and baseline. Baseline for the Extension Period was defined as non-missing assessment in Run-in period prior to the first dose of study drug.
Time Frame: Core Phase: Baseline to Weeks 9-12; Extension Period: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Daily number of flushing episodes
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 14 | 8
Daily number of flushing episodes | -0.88 (1.205) | -1.55 (1.784)

10. Secondary Outcome: Number of Participants Achieving Clinically Meaningful Symptom Reduction in the Core Phase
Description: Clinically meaningful symptom reduction was defined as either: a) an average of < 4 bowel movements per day over 15 consecutive days, b) a 50% reduction from baseline in the number of bowel movements, c) a positive response to the question regarding adequate relief, or d) a 50% reduction from baseline in the number of daily flushing episodes.
Time Frame: Baseline to Week 12
Population: EFAS included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Telotristat Etiprate- Core Phase
Number analyzed (Participants) | 15
Participants | 14

11. Secondary Outcome: Change From Baseline in Urinary 5-Hydroxyindoleacetic Acid (HIAA) Levels
Description: Urinary 5-HIAA (u5-HIAA) is a standard test used in clinical practice to assess the neuroendocrine tumor (NET) activity and is collected as a 24-hour urine specimen. The change from baseline value for the Extension Period was calculated as the difference between mean change in 5-HIAA of the post-baseline interval (Weeks 20 to 21) and baseline. A negative change from baseline indicates improvement. Baseline for the Extension Period was defined as non-missing assessment in Run-in period prior to the first dose of study drug.
Time Frame: Core Phase: Baseline to Week 12; Extension Period: Baseline to Weeks 20-21
Population: Pharmacodynamic (PD) analysis set included all participants who had received at least 1 dose of study drug, had a valid baseline PD assessment, and at least 1 valid post-baseline PD assessment (whole blood 5-HT or u5-HIAA) in Core Phase and Extension Period.
Measure: Mean (Standard Deviation); unit: mg/24 hours
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
Number analyzed (Participants) | 8 | 6
mg/24 hours | -97.26 (164.995) | -65.02 (119.350)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 12 weeks in the Core Phase, up to 124 weeks in the Extension Period and up to 2 weeks in the Follow-up Period
Arm/Group | Telotristat Etiprate- Core Phase | Telotristat Etiprate- Extension Period
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/11
Serious Adverse Events (participants affected / at risk) | 3/15 | 7/11
Other Adverse Events (participants affected / at risk) | 15/15 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telotristat Etiprate- Core Phase (N=15) | Telotristat Etiprate- Extension Period (N=11)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Cardiac operation (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
Therapeutic embolisation (Surgical and medical procedures) | 0 | 2
Carcinoid syndrome (Endocrine disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid heart disease (Cardiac disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telotristat Etiprate- Core Phase (N=15) | Telotristat Etiprate- Extension Period (N=11)
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Carcinoid syndrome (Endocrine disorders) | 0 | 2
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 4 | 1
Lethargy (Nervous system disorders) | 2 | 1
Hypertension (Vascular disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 2
Chest pain (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 3
Oedema peripheral (General disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 3
Carcinoid heart disease (Cardiac disorders) | 0 | 2
Weight decreased (Investigations) | 1 | 2
Migraine (Nervous system disorders) | 1 | 0
Orthostatic intolerance (Nervous system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infected bites (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 1
Blood chromogranin A increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Vitamin D decreased (Investigations) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Flushing (Vascular disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Brunner's gland hyperplasia (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Post embolisation syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Therapeutic embolisation (Surgical and medical procedures) | 0 | 2
Cardiac operation (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.